CLINICAL TRIAL: NCT05972291
Title: Mechanisms of Gulf War Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLD-006-22F; I01CX001477 (NIH)
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Gulf War Illness; Irritable Bowel Syndrome; Gastrointestinal Symptoms
Keywords: gastrointestinal; irritable bowel syndrome; glutamine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: In this study, the investigators will conduct a randomized, double-blind, placebo-controlled clinical trial studying glutamine 5 grams orally three times a day compared to a placebo 5 grams orally three times a day for 12 weeks in 80 Veterans with GWI and GI symptoms. This study will also look at Veterans that have chronic GI symptoms and do not have GWI. The Symptom Severity Scale and intestinal permeability will be measured at baseline, 4, 8, and 12 weeks.
Who Masked: Participant
Masking Description: Each person in this study will receive either glutamine or whey powder to mix in with water. This is done by a random assignment using a computer program for "yes" or "no". All odd numbers of participants will undergo the random choice of the computer program. All even number participants will get the opposite treatment of the previous odd number participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Glutamine (Experimental): You will be asked to consume 5 grams of glutamine three times a day for 12 weeks. At week four, you will be asked to return to the CRC to be assessed, and then to return every four weeks until week 12, which will be the conclusion of the study.
  Interventions: Dietary Supplement: Oral Glutamine
- Whey Protein Powder (Placebo Comparator): You will be asked to consume 5 grams of whey protein powder three times a day for 12 weeks. At week four, you will be asked to return to the CRC to be assessed, and then to return every four weeks until week 12, which will be the conclusion of the study.
  Interventions: Other: Control Arm

INTERVENTIONS:
Dietary Supplement: Oral Glutamine — You will receive an unmarked packet with either glutamine or whey protein powder. Once the packet is opened, the powder should be mixed completely with 8 oz of water. You should completely drink this mixture within 10 minutes. You will consume one packet three times a day for 12 weeks. One packet 30 minutes before breakfast, one packet 30 minutes before lunch, and one packet 30 minutes before the evening meal.
  Arms: Oral Glutamine
Other: Control Arm — You will receive an unmarked packet with either glutamine or whey protein powder. Once the packet is opened, the powder should be mixed completely with 8 oz of water. You should completely drink this mixture within 10 minutes. You will consume one packet three times a day for 12 weeks. One packet 30 minutes before breakfast, one packet 30 minutes before lunch, and one packet 30 minutes before the evening meal.
  Arms: Whey Protein Powder

SUMMARY:
Many veterans with Gulf War Illness developed chronic gastrointestinal symptoms during their deployment to the Persian Gulf. The pathophysiologic mechanisms of these chronic gastrointestinal symptoms are not well understood but cause significant morbidity in veterans. Our proposed studies will provide an innovative and novel treatment trial for chronic gastrointestinal symptoms in veterans with Gulf War Illness that were deployed into war zones. Given that there are currently no specific treatments for these disorders, and that current symptomatic approaches are far from ideal, proof of principle of our trial would be an extremely important advance as it would not only have a beneficial impact on the health of many thousands of our veterans, but also it would substantially reduce the many negative economic effects of this ailment on the VA Health Care System.

DETAILED DESCRIPTION:
Since 2001, more than 2.2 million US veterans have served in Operation Enduring Freedom (OEF) in Afghanistan and Operation Iraqi Freedom (OIF) in Iraq. The Gulf Registry of the VA Environmental Epidemiology Service identified the majority of these veterans as having chronic health complaints of undetermined etiology. Among the symptoms most frequently reported by veterans with Gulf War Illness (GWI) were chronic fatigue, frequent or persistent headache, frequent or persistent muscle or joint pain, and gastrointestinal (GI) symptoms. GI symptoms (e.g., diarrhea, bloating, and abdominal pain) reported by these veterans accounted for most complaints. Indeed, up to 33% of veterans with GWI suffer from chronic GI symptoms.

The investigators have shown that veterans with GWI and GI symptoms have increased intestinal permeability that drives GI symptoms (Zhang et al., 2019). Our research group recently completed a clinical trial demonstrating the effectiveness of oral glutamine supplementation in diarrhea-predominant IBS patients with increased intestinal permeability (Zhou et al., 2019). The investigators now have obtained preliminary evidence that oral glutamine supplementation may restore intestinal permeability in veterans with GWI and GI symptoms. Based on these new findings, the investigators hypothesize that oral glutamine supplementation will improve the Symptom Severity Scale and restore intestinal permeability in veterans with GWI and chronic GI symptoms. The investigators propose to conduct a randomized, double-blind, placebo-controlled clinical trial studying oral glutamine supplementation compared to placebo in veterans with GWI and GI symptoms.

The human GI tract is the major site of glutamine utilization in the body. Glutamine is a major energy source for rapidly dividing intestinal mucosal cells of the digestive tract. Glutamine helps to protect the lining of the GI tract. Its depletion results in epithelial atrophy and a subsequent increase in intestinal permeability. Glutamine supplementation has been shown to decrease bacterial translocation and intestinal permeability after intestinal injury. Glutamine supplementation has also been shown to decrease intestinal permeability and improve GI function in patients with Crohn's disease, advanced esophageal cancer, or metastatic cancer undergoing radio chemotherapy. There are no published studies to date to support the use of glutamine for veterans with GWI and chronic GI symptoms.

However, given our published studies, preliminary data demonstrating restoration of intestinal permeability with oral glutamine therapy, and the mechanisms of action of glutamine on the GI tract, research testing whether oral glutamine is an effective therapy in veterans with GWI is needed. Given that there are no effective treatments for these veterans and that current treatment approaches are far from ideal, this proposed clinical trial would be extremely important as it would not only have a beneficial impact on the health of many of our veterans, but also it would substantially reduce the negative economic effects on the VA Health Care System.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans 18-65 years old with GWI and chronic GI symptoms (abdominal pain, diarrhea, bloating) that started during their deployment in the Persian Gulf
2. Veterans 18-65 years old with GWI and chronic GI symptoms (abdominal pain, diarrhea, bloating)
3. increased intestinal permeability on the lactulose/mannitol permeability test (ratio >0.07)
4. able and willing to cooperate with the study

Exclusion Criteria:

1. current participation in another research protocol or unable to give informed consent
2. women with a positive urine pregnancy test or breastfeeding
3. history of inflammatory bowel disease, lactose intolerance and/or celiac sprue
4. + hydrogen breath test for bacterial overgrowth
5. + anti-endomysial antibody titer
6. use of NSAIDs 2 weeks before or during the study
7. known allergy to glutamine or whey protein
8. abdominal surgery except for removal of gallbladder, uterus, or appendix >6 months prior to entry into the study
9. Abnormal serum BUN and/or creatinine
10. Mannitol recovery out of the normal range of 5-25 U/g
11. history of kidney disease
12. allergies to monosodium glutamate
13. current use of anti-seizure medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine if oral glutamine supplementation will improve the Symptom Severity Scale in Veterans with GWI and chronic GI Symptoms. | 3 years
  It's anticipated that veterans with GWI and GI symptoms will show a significant reduction, compared to placebo, in their chronic GI symptoms as reflected by their Symptom Severity Scale Score following glutamine therapy. For each participating subject, the Symptom Severity Scale score will be measured at baseline, and at 4, 8, and 12 weeks after the start of treatment. The investigators will have Symptom Severity Scale scores at 5 time points in each group (glutamine, placebo). These will be explored graphically with time course plots. At each time point, for Symptom Severity Scale scores, the investigators will also calculate descriptive statistics including mean and standard deviation, as well as median, median absolute deviation and inter-quartile range if the distribution of data is skewed. Box plots will be used to graphically demonstrate the distribution of Symptom Severity Scale scores at each time point. This will be done for both the glutamine and the placebo groups.
To determine if oral glutamine supplementation will restore intestinal permeability in Veterans with GWI. | 3 years
  Following our recent findings, we expect >75% of veterans will restore normal intestinal permeability, while in the placebo group, this percentage is ~6%. One sample one sided proportion test (PROC FREQ in SAS) will be used to test whether the proportion of restoration is >75% in each treatment group (glutamine supplementation or placebo) and two sample one sided proportion tests (PROC FREQ in SAS) to compare the difference between the two groups. To examine the association between the Symptom Severity Scale Score and restoration of normal intestinal permeability, Pearson's correlations between the Symptom Severity Scale and intestinal permeability will be calculated at baseline, and at 4, 8, and 12 weeks after the start of treatment, for both oral glutamine and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: QiQi Zhou, MD PhD, Principal Investigator — Memphis VA Medical Center, Memphis, TN; George N Verne, Principal Investigator — Memphis VA Medical Center, Memphis, TN
Locations (1):
- Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No